CLINICAL TRIAL: NCT07332858
Title: First-in-Human Expanded Cohort Study of Intrapleural Administration of TolueneSulfonamide in Patients With Malignant Pleural Effusion
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gang Hou (Other)
Collaborators: The Second Affiliated Hospital of Harbin Medical University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Anhui Chest Hospital (Other)
Responsible Party: Sponsor-Investigator, Gang Hou, Chief Physician, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-HX-183
Record Dates: First submitted 2025-12-19; First posted 2026-01-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Malignant Pleural Effusions (Mpe); Non Small Cell Lung Cancer
Keywords: Malignant Pleural Effusion; Para-toluenesulfonamide
MeSH Terms: conditions — Pleural Effusion, Malignant; Myeloproliferative Disorder, Chronic, with Eosinophilia; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: This study consists of two parts. Part 1 is a first-in-human study enrolling 15 patients with malignant pleural effusion (MPE) to assess the safety of intrapleural PTS. Part 2 will enroll 90 patients with MPE and, after safety is confirmed, randomize them 2:1 to receive PTS plus catheter drainage or normal saline plus catheter drainage. Treatment is given in weekly cycles with dosing on Days 1, 3, and 5. Pleural effusion is drained before each dose, followed by intrapleural administration and catheter clamping. After treatment, standard drainage and supportive care are continued.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrapleural PTS injection plus catheter drainage group (Experimental): PTS Administration (One Treatment Cycle):
  One treatment cycle is defined as one week. PTS is administered three times per week on Days 1, 3, and 5. Prior to each administration, pleural effusion is drained as completely as possible until no further fluid can be obtained. The study drug is then administered via the indwelling drainage catheter, followed by an additional flush of 20 mL of normal saline. The drainage catheter is clamped for at least 24 hours after administration.
  After each injection, patients are instructed to maintain prone, lateral, and supine positions for approximately 30 minutes each to facilitate even distribution of the drug within the pleural cavity. During the same treatment cycle, the drainage catheter remains clamped until the next scheduled administration. After completion of treatment, catheter drainage and standard care are continued.
  Interventions: Drug: Intrapleural administration of TolueneSulfonamide
- catheter drainage alone group (Placebo Comparator): Normal Saline Administration (One Treatment Cycle):
  One treatment cycle is defined as one week. Normal saline is administered three times per week on Days 1, 3, and 5. Prior to each administration, pleural effusion is drained as completely as possible until no further fluid can be obtained. Normal saline is then administered via the indwelling drainage catheter, followed by an additional flush of 20 mL of normal saline. The drainage catheter is clamped for at least 24 hours after administration.
  After each administration, patients are instructed to maintain prone, lateral, and supine positions for approximately 30 minutes each. During the same treatment cycle, the drainage catheter remains clamped until the next scheduled administration. After completion of treatment, catheter drainage and standard care are continued.
  Interventions: Drug: Intrapleural administration of normal saline injection

INTERVENTIONS:
Drug: Intrapleural administration of TolueneSulfonamide — PTS Administration (One Treatment Cycle):
  One treatment cycle is defined as one week. PTS is administered three times per week on Days 1, 3, and 5. Prior to each administration, pleural effusion is drained as completely as possible until no further fluid can be obtained. The study drug is then administered via the indwelling drainage catheter, followed by an additional flush of 20 mL of normal saline. The drainage catheter is clamped for at least 24 hours after administration.
  After each injection, patients are instructed to maintain prone, lateral, and supine positions for approximately 30 minutes each to facilitate even distribution of the drug within the pleural cavity. During the same treatment cycle, the drainage catheter remains clamped until the next scheduled administration. After completion of treatment, catheter drainage and standard care are continued.
  Arms: Intrapleural PTS injection plus catheter drainage group
Drug: Intrapleural administration of normal saline injection — Normal Saline Administration (One Treatment Cycle):
  One treatment cycle is defined as one week. Normal saline is administered three times per week on Days 1, 3, and 5. Prior to each administration, pleural effusion is drained as completely as possible until no further fluid can be obtained. Normal saline is then administered via the indwelling drainage catheter, followed by an additional flush of 20 mL of normal saline. The drainage catheter is clamped for at least 24 hours after administration.
  After each administration, patients are instructed to maintain prone, lateral, and supine positions for approximately 30 minutes each. During the same treatment cycle, the drainage catheter remains clamped until the next scheduled administration. After completion of treatment, catheter drainage and standard care are continued.
  Arms: catheter drainage alone group

SUMMARY:
This study aims to evaluate the safety of intrapleural injection of TolueneSulfonamide in patients with malignant pleural effusion and to explore its potential effectiveness.

DETAILED DESCRIPTION:
This study is a first-in-human (FIM) expansion cohort study designed to evaluate the safety and clinical activity of intrapleural injection of PTS in patients with malignant pleural effusion (MPE). Patients with MPE will be prospectively enrolled, and the study will be conducted in two parts: a safety and dose-exploration phase of intrapleural PTS administration (Part 1, P1), followed by an efficacy evaluation phase of intrapleural PTS for the treatment of MPE (Part 2, P2). Part 2 will be initiated after the safety of PTS has been established in Part 1.

Part 1 is designed as a prospective, single-arm, open-label study. Part 2 is designed as a prospective, multicenter, double-blind, randomized controlled trial with two groups: an experimental group and a control group. The experimental group will receive catheter drainage plus intrapleural PTS injection, while the control group will receive catheter drainage plus intrapleural normal saline injection.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years (inclusive) at the time of signing the informed consent form.
2. Histologically or cytologically confirmed malignant pleural effusion, with the primary tumor diagnosed as non-small cell lung cancer (NSCLC).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2, with an expected survival of at least 3 months.
4. Presence of dyspnea symptoms.
5. No prior local thoracic treatment within 1 month before enrollment, including intrapleural drug administration or thoracic radiotherapy (diagnostic thoracentesis is permitted).
6. Except for the subject's current stable systemic anti-tumor therapy, any other ongoing tumor-related treatments must be suspended or discontinued after evaluation by the investigator to ensure they do not interfere with the assessment of PTS treatment.
7. Fully understands the study objectives and procedures, agrees to participate in the study, and provides written informed consent.

Exclusion Criteria:

1. History of allergy or hypersensitivity to PTS or any of its excipients.
2. Presence of uncontrolled intrapleural infection or severe loculated pleural effusion that is difficult to manage.
3. Participation in another interventional clinical study within 3 months prior to enrollment (diagnostic studies are excluded).
4. Severe organ dysfunction, including but not limited to coagulation disorders, congestive heart failure, malignant arrhythmias, coronary artery disease requiring long-term medication, valvular heart disease, myocardial infarction, or refractory hypertension; severe cardiac, hepatic, or renal insufficiency, or active bleeding or thrombotic risk.
5. Presence of uncontrolled infectious wounds.
6. Pregnant or breastfeeding women.
7. Any other condition that, in the investigator's judgment, makes the subject unsuitable for participation in this study.
8. Criteria for withdrawal from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 4 weeks, 12 weeks, 6 months, and 12 months after treatment completion
  Objective Response Rate (ORR) is defined as the proportion of patients achieving complete response (CR) or partial response (PR) among all enrolled patients, calculated as (CR + PR) / total number of patients × 100%, based on WHO criteria and assessed by imaging methods (ultrasound or computed tomography).

SECONDARY OUTCOMES:
Percentage Change in Pleural Effusion Volume | Baseline; after one treatment cycle (each cycle is 7 days); and at 4 weeks, 12 weeks, 6 months, and 12 months of follow-up
  The rate of change in pleural effusion volume is calculated as (baseline pleural effusion volume - post-treatment pleural effusion volume) / baseline pleural effusion volume, with pleural effusion volume assessed by ultrasound and computed tomography (CT)
Overall Survival (OS) | through study completion, an average of 1 year
  the time from enrollment to death from any cause
Incidence of Grade ≥3 treatment-emergent adverse events | through study completion, an average of 1 year
  Incidence of Grade ≥3 treatment-emergent adverse events
mMRC Dyspnea Score | At baseline, after one treatment cycle (each cycle is 7 days), and at 4 weeks, 12 weeks, 6 months, and 12 months during follow-up
  Dyspnea will be assessed using the modified Medical Research Council (mMRC) Dyspnea Scale.
Quality of Life score | At baseline, after one treatment cycle (each cycle is 7 days), and at 4 weeks, 12 weeks, 6 months, and 12 months during follow-up
  Quality of life will be assessed using the EORTC QLQ-C30 (core questionnaire) together with the QLQ-LC13 (lung cancer-specific module), or the EuroQol five-dimension questionnaire (EQ-5D).

CONTACTS AND LOCATIONS:
Overall Officials: Gang Hou, PhD, Study Director — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Guan WJ, Li SY, Zhong NS. Effects of para-toluenesulfonamide intratumoral injection on pulmonary adenoid cystic carcinoma complicating with severe central airway obstruction: a 5-year follow-up study. J Thorac Dis. 2018 Apr;10(4):2448-2455. doi: 10.21037/jtd.2018.03.70. PMID 29850151
- [Background] Li SY, Li Q, Guan WJ, Huang J, Yang HP, Wu GM, Jin FG, Hu CP, Chen LA, Xu GL, Liu SZ, Wu CG, Han BH, Xiang Y, Zhao JP, Wang J, Zhou X, Li HP, Zhong NS. Effects of para-toluenesulfonamide intratumoral injection on non-small cell lung carcinoma with severe central airway obstruction: A multi-center, non-randomized, single-arm, open-label trial. Lung Cancer. 2016 Aug;98:43-50. doi: 10.1016/j.lungcan.2016.05.012. Epub 2016 May 17. PMID 27393505
- [Background] Xu YF, Chen YR, Bu FL, Huang YB, Sun YX, Li CY, Sellick J, Liu JP, Qin DM, Liu ZL. Chinese herbal injections versus intrapleural cisplatin for lung cancer patients with malignant pleural effusion: A Bayesian network meta-analysis of randomized controlled trials. Front Oncol. 2022 Sep 20;12:942941. doi: 10.3389/fonc.2022.942941. eCollection 2022. PMID 36203451
- [Background] Dong X, Huang Y, Yi T, Hu C, Gao Q, Chen Y, Zhang J, Chen J, Liu L, Meng R, Zhang S, Dai X, Fei S, Jin Y, Yin P, Hu Y, Wu G. Intrapleural infusion of tumor cell-derived microparticles packaging methotrexate or saline combined with pemetrexed-cisplatin chemotherapy for the treatment of malignant pleural effusion in advanced non-squamous non-small cell lung cancer: A double-blind, randomized, placebo-controlled study. Front Immunol. 2022 Oct 5;13:1002938. doi: 10.3389/fimmu.2022.1002938. eCollection 2022. PMID 36275698
- [Background] Feller-Kopman DJ, Reddy CB, DeCamp MM, Diekemper RL, Gould MK, Henry T, Iyer NP, Lee YCG, Lewis SZ, Maskell NA, Rahman NM, Sterman DH, Wahidi MM, Balekian AA. Management of Malignant Pleural Effusions. An Official ATS/STS/STR Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Oct 1;198(7):839-849. doi: 10.1164/rccm.201807-1415ST. PMID 30272503
- [Background] Porcel JM, Cordovilla R, Tazi-Mezalek R, Barrios-Barreto D, Perez-Pallares J, Novais E Bastos H, Martinez-Tomas R, Flandes-Aldeyturriaga J, Cases-Viedma E, Recalde B, Botana-Rial M. Efficacy and Safety of Indwelling Catheter for Malignant Pleural Effusions Related to Timing of Cancer Therapy: A Systematic Review. Arch Bronconeumol. 2023 Sep;59(9):566-574. doi: 10.1016/j.arbres.2023.06.007. Epub 2023 Jun 23. English, Spanish. PMID 37429748
- [Background] 北京肿瘤学会临床研究专委会，中国医院协会肿瘤医院分会，王书航，等。恶性胸腔积液干预性临床研究设计专家共识[J]. 中华肿瘤防治杂志, 2025,32(8): 455-461.
- [Background] Kumar A, Xu B, Srinivasan D, Potter AL, Raman V, Lanuti M, Yang CJ, Auchincloss HG. Long-Term Survival of American Joint Committee on Cancer 8th Edition Staging Descriptors for Clinical M1a Non-Small Cell Lung Cancer. Chest. 2024 Mar;165(3):725-737. doi: 10.1016/j.chest.2023.07.4220. Epub 2023 Aug 5. PMID 37544427